CLINICAL TRIAL: NCT00481026
Title: A Double Blind Sham Controlled Trial of tDCS in Treating Schizophrenia and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11707
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia; Major Depression
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Sham Comparator): Placebo tDCS
  Interventions: Device: transcranial direct current stimulation (tDCS)
- active tDCS (Active Comparator): active tDCS
  Interventions: Device: active tDCS

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS
  Arms: Placebo
Device: active tDCS — Active tDCS
  Arms: active tDCS

SUMMARY:
The project will investigate the use of a novel technique, transcranial direct current stimulation (tDCS) in the treatment of patients with schizophrenia and patients with depression. tDCS involves the application of an extremely weak continuous electrical current to the brain through the placement of anode and a cathode on the scalp. The electrical current is generally completely imperceptible after initial period of tingling which takes about 30 seconds. Stimulation under the anode appears to increase brain activity where as stimulation under the cathode has the opposite effect. This research plan involves two clinical trials:

1. A study using tDCS to treat both the positive and negative symptoms of schizophrenia. The negative symptoms of schizophrenia such as lack of motivation and energy appear to arise due to a lack of activity in frontal brain areas. Positive symptoms such as hallucinations and confused thoughts may arise through over activity of brain areas more on the side and towards the back of the brain called the temporal cortex. We plan to apply tDCS such that it can simultaneously increased activity in these frontal brain areas and reduce activity over temporal cortex. We will compare active stimulation to a placebo condition which involves turning the stimulator off after 30 seconds. The capacity to target multiple symptom clusters is unique with this type of brain stimulation.
2. The study using tDCS in treatment resistant depression builds on a work with transcranial magnetic stimulation (TMS). TMS techniques in depression seem to work which increased left frontal brain activity or decrease right frontal brain activity. tDCS will be used to do the same thing with the anode used to increase left-sided brain activity and the cathode used to simultaneously decreased right-sided brain activity.

tDCS is potentially a better tolerated procedure than TMS and does not appear to have the same risk of seizure induction. Importantly, the equipment is quite inexpensive and this may prove to be an extremely safe and effective low-cost treatment for psychiatric disorders in Third World countries.

DETAILED DESCRIPTION:
TREATMENT OF MAJOR DEPRESSION USING TRANSCRANIAL DIRECT CURRENT STIMULATION

Rationale:

Depression and tDCS Major depression is a disorder with major clinical and economic significance locally and internationally. It is a disorder of high prevalence and results in substantial disease burden and health-care costs. Critically, a significant percentage of patients, usually estimated at around 30%, fail to respond to standard treatments (Fitzgerald 2003). Techniques such as repetitive transcranial magnetic stimulation (rTMS) are being investigated widely for the treatment of this disorder with considerable success in recent years (Fitzgerald, Benitez et al. 2006)(Hasey 2001). However, TMS equipment is expensive and requires specialist application. Additionally, TMS is associated with some side-effects. Given that depression occurs in all cultures and countries, there would be considerable value in developing a low-cost, non-invasive technique that can be applied in a wide variety of settings, including in the Third World.

RTMS based treatments for depression are based on an understanding that there are abnormalities in activity in frontal brain regions in this disorder (George, Ketter et al. 1994; Fitzgerald, Brown et al. 2003; Speer, Kimbrell et al. 2000). High-frequency stimulation which increases brain activity is usually applied to the left prefrontal cortex in a way that increases activity, although previous literature is somewhat inconsistent. In contrast, low-frequency stimulation which decreases brain activity is applied to the right prefrontal cortex to reduce activity in this region. Both these techniques have therapeutic efficacy (Fitzgerald, Brown et al. 2003). Recent studies, including those conducted by this research group, suggest that a combination of these two approaches is also effective; potentially more effective than either one used independently (Garcia-Toro, Salva et al. 2006; Fitzgerald, 2006).

Transcranial direct current stimulation (tDCS) is a novel, non-invasive and non-convulsive technique for altering brain function (Ardolino, Bossi et al. 2005). It involves the application of a small current (usually 1 to 2 mA) between an anodal and cathodal electrode placed on the scalp (Miranda, Lomarev et al. 2006). Typically, an increase in neuronal excitability occurs under the anode, and a decrease under the cathode, probably through respective depolarisation and hyperpolarisation of neurons (Miranda, Lomarev et al. 2006). It has been shown to be safe in a number of experimental and clinical trials (Fregni, Boggio et al. 2005; Fregni, Boggio et al. 2005; Fregni, Boggio et al. 2006; Fregni, Boggio et al. 2006; Nitsche, Liebetanz et al. 2003; Lang, Nitsche et al. 2004; Boggio, Castro et al. 2006).

Most of the research with tDCS has investigated its use in modifying cognitive functions in experimental neuropsychology. However there is an increasing use of this technique in therapeutic trials for disorders such as chronic pain, tinnitus and motor impairment post-stroke (Fregni, Boggio et al. 2005; Fregni, Boggio et al. 2006). Research has also begun on tDCS in the treatment of depression (Nitsche 2002; Fregni, Boggio et al. 2006). In the first of these studies patients were randomised to active or sham stimulation (Fregni, Boggio et al. 2006). Anodal stimulation was applied to the left prefrontal cortex. This resulted in statistically significant improvement in depressive symtomology, relative to the sham condition. As the sensation produced by tDCS usually disappears completely after 30 seconds, the sham used in this study involves turning the device on for 30 seconds and then turning it off. A second study by the same group including 30 patients has been submitted for publication. It also shows statistically significant antidepressant effects on the active treatment group, relative to sham stimulation. Importantly, no substantial side-effects have been reported in either of these two clinical trials (Fregni, Boggio et al. 2006).

Both of these two studies in depression have used anodal stimulation applied to the left prefrontal cortex. The cathode was placed in a position over the left eye and was proposed not to have contributed to the antidepressant efficacy of the stimulation. We propose a slightly different protocol involving anodal stimulation to the left prefrontal cortex and the placement of the cathode over the right prefrontal cortex. This should ensure activating stimulation on the left and deactivating stimulation on the right quite similar to the sequential bilateral rTMS techniques that we have been testing. There is no reason to presume that this should be associated with any greater rate of side-effects, but may enhance therapeutic efficacy.

General Study Design: The proposed study will be a randomized, double blind, placebo-controlled (i.e., sham tDCS), longitudinal, treatment outcome trial. Individuals with depression will be randomized to 1 of 2 treatment conditions. These will be:

1. Active 2mA transcranial direct current stimulation (tDCS): in this condition, 1 stimulator will be used with anodal stimulation to the left prefrontal cortex and cathodal stimulation to the right prefrontal cortex. The placement of anodal stimulation is proposed to enhance activity in the left frontal cortex; and the cathode aims to reduce activity in the right prefrontal cortex.
2. Sham treatment: the system will be set up as for condition one but the stimulated will be turned off after 30 seconds.

A total of 15 treatments will be administered to all participants over 3 weeks (one per working day). Individuals will be randomized on a computer-generated list with the information stored on a central computer such that only the treating physician will be aware of the treatment allocation of the patients. It is anticipated that stratified randomization of the sample according to potentially clinically significant variables such as age, sex, illness and treatment duration would dramatically increase the required sample size and is beyond the scope of this study. Therefore, we have chosen not to do so. Nonetheless, based on descriptive statistics, multiple linear regression will be performed to adjust for significant clinical predictors. Clinical raters and patients will be blind to the treatment condition. The following primary hypotheses will be tested.

* Hypothesis 1: Active tDCS will improve depressive symptomology to a significantly greater degree than sham treatment.
* Hypothesis 2: Active tDCS will be well tolerated and free of major side effects.

Subjects: 50 patients with depression will be recruited to participate in the study.

* Participants will be included if they: (1) Are competent to consent; (2) have a diagnosis of Major Depression and are currently experiencing a Major Depressive Episode as confirmed by the Structure Clinical Interview for the DSM-IV (SCID-IV); (3) are treatment resistant, defined as a failure to achieve a clinical response, or an inability to tolerate, an antidepressant trial of sufficient dose for at least 6 weeks; and (4) are between the ages of 18 and 75. Concomitant medications including: (1) benzodiazepines, (2) mood stabilizers (lithium, valproic acid) (3) antidepressants (including serotonin reuptake inhibitors and tricyclic antidepressants) and anticholinergics will be allowed. Since carbamazepine has been shown to interfere with the effects of anodal tDCS, potential participants taking it will not be suitable for inclusion in the trial.
* Patients will be excluded if they: (1) Have a DSM-IV history of substance abuse or dependence in the last 6 months; (2) Have a concomitant major and unstable medical or neurologic illness; (4) are currently taking carbamazepine; or, (3) are pregnant.
* Finally, patients will be withdrawn from the study if they: (1) withdraw consent; (2) experience significant clinical deterioration; (3) fail to tolerate the procedure; or, (4) develop a serious adverse event. In the event that a patient is withdrawn or drops out of the study, efforts will be made to obtain a final set of clinical, cognitive and neurophysiological measures at the time of withdrawal for a last observation carried forward analysis.

Transcranial direct current stimulation:

Site, Intensity and Frequency: Direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and delivered by a specially developed, battery driven constant current stimulator. The electrodes will be placed over F3 and F4 according to the 10-20 international system for EEG placement. This has been shown to be a relatively accurate method of dorsolateral prefrontal cortex (DLPFC) localisation by neuronavigation methods (Herwig, Padberg et al. 2001), and has been used before in tDCS studies targeting the dorsolateral prefrontal cortex (Fregni, Boggio et al. 2005; Fregni, Boggio et al. 2006).

Safety: tDCS has previously been used in multiple studies in areas such as post-stroke rehabilitation, Parkinson's disease and depression, with no adverse sequelae noted (Fregni, Boggio et al. 2005; Fregni, Boggio et al. 2005; Fregni, Boggio et al. 2006; Fregni, Boggio et al. 2006)(Nitsche, Liebetanz et al. 2003; Lang, Nitsche et al. 2004; Boggio, Castro et al. 2006). The procedure produces a mild tingling sensation initially which has usually completely resolved within 30 seconds.

Sham Condition: Sham stimulation will be made using the same stimulation parameters and at the site of active treatment, but the current will be turned off after 30 seconds. Typically, tDCS induces an itching or tingling sensation for the first 30 seconds of its application, which then fades, making this an appropriate method for blinding.

Course: The primary study will be 3 weeks in duration. Therefore, participants will receive 15 treatments lasting twenty minutes, conducted daily on week days. Patients will be assessed at baseline and 3 weeks and with an abbreviated assessment after the first 7 days of treatment (MADRS only). Patients in the sham group will be offered open label active treatment at the end. Patients who have responded to tDCS will also be followed up post treatment with assessments at up to monthly intervals where possible to assess duration of response. Patients who have achieved a significant response to tDCS may be offered a 'repeat' treatment if requested following symptomatic relapse.

Symptoms: Symptoms of depression will be assesed with the 17-item Hamilton Rating Scale for Depression (HAMD). Other outcome measures will include the Montgomery-Asberg Depression Rating Scale (MADRS), Beck Depression Questionnaire (BDI), Brief Psychiatric Rating Scale (BPRS) and an interview to record the subjective experiences of tDCS and any adverse events.

Cognition: The primary outcome measures will be performance on the forwards and backwards digit span (assessment of verbal working memory) and block spatial span (spatial working memory) tests. In addition, other aspects of prefrontal cognitive functioning will be assessed using the N-back task, Tower of London planning task, FAS verbal fluency task and the trail making task (A &B). These additional task are included to assess whether treatment with rTMS results in specific changes to working memory or broader domains of prefrontal cognitive functioning. In addition, baseline assessment of premorbid intellectual functioning will be conducted using the Wechsler Adult Intelligence Scale - 3rd edition (WAIS-III).

Electroencephalography: Where possible (based on laboratory availability) EEG will be recorded before and after tDCS to assess the effect of tDCS on alpha, beta, delta, theta and gamma power bands using a standard 64 channel Neuroscan EEG system used in many studies by our group.

Analysis We will use a series of repeated measures ANOVA models to assess change in depressive and cogntive symptoms over time between the groups. There is no data on which to base a smaple size calculation: we have planned a larger sample than that used in most rTMS and tDCS trials and will conduct an interim analysis after the recruitment of 20 patients to re-estimate the sample size.

THE TREATMENT OF WORKING MEMORY AND NEGATIVE SYMPTOMS IN PATIENTS WITH SCHIZOPHRENIA WITH TRANSCRANIAL DIRECT CURRENT STIMULATION

Rationale:

Schizophrenia and tDCS

Schizophrenia (SCZ) is a debilitating disease which affects approximately 1% of the population. Measured only in an economic sense, the cost to the Australian government is estimated at 2.25 billion Australian dollars per annum [1]. A significant proportion of the burden carried by individuals with schizophrenia stems from negative symptoms such as social withdrawal and impaired executive functioning. Current treatments for schizophrenia, including new atypical antipsychotic agents, while effective in treating some positive symptoms of schizophrenia, have demonstrated only limited efficacy in treating negative symptoms. There is a need for a new therapeutic option for people with schizophrenia which can treat these aspects of their illness.

Transcranial direct current stimulation (tDCS) is a novel, non-invasive and non-convulsive technique for altering brain function. It involves the application of a small current (usually 1 to 2 mA) between an anodal and cathodal electrode which are placed on the scalp. Typically, an increase in neuronal excitability occurs under the anode, and a decrease under the cathode, probably through depolarisation and hyperpolarisation of neurons, respectively [2]. It has been shown to be safe in a number of experimental and clinical trials [3] and therapeutic benefits have been found in using it in the treatment of depression, pain disorders, tinnitus and motor impairment post stroke [4, 5]. In depression, one study has shown therapeutic effects compared to sham stimulation and the same group have a second positive study of 40 patients currently under review. This clearly shows antidepressant effects of tDCS greater than sham and no side effects. In fact, side effects in previous trials have been limited to a mild transient sensation of itching or tingling underneath the site of the electrodes [4]. Previous studies have shown that transcranial magnetic stimulation (TMS) [6, 7], another technique of neuromodulation, may be effective in treating positive and negative symptoms of schizophrenia. However TMS at the high frequencies required to increase brain activity can be physically uncomfortable due to the induction of scalp muscle twitching and is associated with potential seizure induction. tDCS is considerably cheaper than TMS, at approximately one tenth of the cost, and is associated with fewer side effect so may have a role to play in alleviating some of the disease burden for people who have schizophrenia.

Negative symptoms, prefrontal cortex and short term memory

A number of studies have found an association between negative symptoms including blunted affect and executive functioning cognitive deficits and reduced activation in prefrontal areas, particularly the left prefrontal cortex. [8-14]. Biltaeral dorsolateral left prefrontal cortex dysfunction has been associated with short term memory deficits in schizophrenia [15]. Application of tDCS to the left prefrontal cortex has been shown to improve short term memory [16]. As such, treatment with tDCS would appear to have the potential to improve short term memory deficits in individuals with schizophrenia, and it also may have a positive impact on their negative symptom.

General Study Design: The proposed study will be a randomized, double blind, placebo-controlled (i.e., sham tDCS), longitudinal, treatment outcome trial. Individuals with SCZ will be randomized to 1 of 2 treatment conditions. These will be:

1. Bilateral 2mA transcranial direct current stimulation (tDCS): in this condition, 2 stimulators will be used with anodal stimulation to the prefrontal cortex and cathodal stimulation to temporoparietal cortex (TP3 EEG site). The placement of anodal stimulation is proposed to enhance activity in bilateral frontal cortex and potentially improve negative and cognitive symptoms. Bilateral rTMS designed to reduce cortical activity appears to improve negative symptoms [17].

   The cathodes, which should reduced cortical activity, are being placed over temporoparietal cortex: this site is proposed to be hyper-active in positive symptoms of schizophrenia including hallucinations and possibly delusions and thought disorder [18-22]. rTMS than reduces activity (analogous to cathodal stimulation) has been shown to reduce these symptoms, especially hallucinations (for example [1, 23, 24]).

   Thus, with these electrode arrangements, we anticipate the potential treatment of both positive and cognitive / negative symptoms simultaneously. This would not be possible with other brain stimulation techniques that only target one site (e.g. rTMS).
2. Sham treatment

A total of 15 treatments will be administered to all participants over 3 weeks (one per working day). Individuals will be randomized on a computer-generated list with the information stored on a central computer such that only the treating physician will be aware of the treatment allocation of the patients. It is anticipated that stratified randomization of the sample according to potentially clinically significant variables such as age, sex, illness and treatment duration would dramatically increase the required sample size and is beyond the scope of this study. Therefore, we have chosen not to do so. Nonetheless, based on descriptive statistics, multiple linear regression will be performed to adjust for significant clinical predictors. Clinical raters and patients will be blind to the treatment condition. The following primary hypotheses will be tested.

* Hypotheses 1: Bilateral tDCS will improve working memory in subjects with schizophrenia
* Hypothesis 2: Bilateral tDCS will reduce negative symptoms in subjects with schizophrenia.
* Hypothesis 3: Bilateral tDCS will reduce positive symptoms in subjects with schizophrenia.

Subjects: 50 patients with SCZ will be recruited to participate in the study.

* Participants will be included if they: (1) Are voluntary and competent to consent; (2) have a diagnosis of Schizophrenia or Schizoaffective Disorder as confirmed by the Structure Clinical Interview for the DSM-IV (SCID-IV) (3) have persistent positive and negative symptoms despite having trialled, or being currently medicated, with antipsychotic medication; and (4) are between the ages of 18 and 65. Concomitant medications including: (1) benzodiazepines, (2) mood stabilizers (lithium, valproic acid) (3) antidepressants (including serotonin reuptake inhibitors and tricyclic antidepressants) and anticholinergics will be allowed. Since carbamazepine has been shown to interfere with the effects of anodal tDCS, potential participants taking it will not be suitable for inclusion in the trial.
* Patients will be excluded if they: (1) Have a DSM-IV history of substance abuse or dependence in the last 6 months; (2) Have a concomitant major and unstable medical or neurologic illness or have had a history of seizures; (4) are currently taking carbamazepine; or, (3) are pregnant.
* Finally, patients will be withdrawn from the study if they: (1) withdraw consent; (2) experience significant clinical deterioration; (3) fail to tolerate the procedure; or, (4) develop a serious adverse event (e.g., seizure activity, active suicidal ideation). In the event that a patient is withdrawn or drops out of the study, efforts will be made to obtain a final set of clinical, cognitive and neurophysiological measures at the time of withdrawal for a last observation carried forward analysis.

No restriction on inclusion will be made based on baseline WM performance. This will allow us to study a broad range of the spectrum of WM performance as well as the effects of tDCS on performance that is potentially normal as well as impaired. Data available for memory impairment in general suggests that ~80% of patients with SCZ will perform below the median within a sample of patients and controls [25] suggesting it is likely that in an unselected sample of patients with SCZ, we are highly likely to see a significant majority with WM performance below the mean for control subjects.

Transcranial direct current stimulation:

Site, Intensity and Frequency: Direct current will be transferred with a pair of saline soaked sponge electrodes (contact area 5 x 7cm), and delivered by a specially developed, battery driven constant current stimulator. The anode electrode will be placed over F3 according to the 10-20 international system for EEG placement. This has been shown to be a relatively accurate method of dorsolateral prefrontal cortex (DLPFC) localisation by neuronavigation methods [26], and has been used before in tDCS studies targeting the dorsolateral prefrontal cortex [4, 16]. The cathodal electrode will be placed over the left temporal area (TP3 EEG site). Twenty minutes of 2mA stimulation will be applied in a regime previously shown to enhance working memory in a population with Parkinson's disease at a level of 2mA [4]. The same procedure will also be applied on the right side.

Safety: tDCS has previously been used in multiple studies in areas such as post-stroke rehabilitation, Parkinson's disease and depression, with no adverse sequelae noted. [4, 5, 16, 27]. The procedure produces a mild tingling sensation initially which has usually completely resolved within 30 seconds.

Sham Condition: Sham stimulation will be made using the same stimulation parameters and at the site of active treatment, but the current will be turned off after 30 seconds. Typically, tDCS induces an itching or tingling sensation for the first 30 seconds of its application, which then fades, making this an appropriate method for blinding [5].

Course: The primary study will be 3 weeks in duration. Therefore, participants will receive 15 treatments lasting twenty minutes, conducted daily on week days. Patients will be assessed at baseline and 3 weeks and with an abbreviated assessment after the first 7 days of treatment (PANSS only). Patients in the sham group will be offered open label active treatment at the end. Patients who have responded to tDCS will also be followed up post treatment with assessments at up to monthly intervals where possible to assess duration of response. Patients who have achieved a significant response to tDCS may be offered a 'repeat' treatment if requested following symptomatic relapse.

Cognition: The primary outcome measures will be performance on the forwards and backwards digit span (assessment of verbal working memory) and block spatial span (spatial working memory) tests. In addition, other aspects of prefrontal cognitive functioning will be assessed using the N-back task, Tower of London planning task, FAS verbal fluency task and the trail making task (A &B). These additional task are included to assess whether treatment with rTMS results in specific changes to working memory or broader domains of prefrontal cognitive functioning. In addition, baseline assessment of premorbid intellectual functioning will be conducted using the Wechsler Adult Intelligence Scale - 3rd edition (WAIS-III)([28]).

Symptoms: Symptoms of schizophrenia will be assesed with the Positive and Negative Symptom Scale (PANSS) [29]. In addition, as prefrontal tDCS may well modify negative symptoms, these will be assessed in more detail with the Scale for the Assessment of Negative Symptoms (SANS) [30]. We will allow for the capacity to control for effects on mood of prefrontal rTMS by assessing depression with the Calgary Depression Scale [31].

Electroencephalography: Where possible (based on laboratory availability) EEG will be recorded before and after tDCS to assess the effect of tDCS on alpha, beta, delta, theta and gamma power bands using a standard 64 channel Neuroscan EEG system used in many studies by our group.

Analysis We will use a series of repeated measures ANOVA models to assess change in positive, negative and cogntive symptoms over time between the groups. There is no data on which to base a smaple size calculation: we have planned a larger sample than that used in most rTMS and tDCS trials and will conduct an interim analysis after the recruitment of 20 patients to re-estimate the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Participants will be included if they:

  1. Are voluntary and competent to consent;
  2. Have a diagnosis of Schizophrenia or Schizoaffective Disorder as confirmed by the Structure Clinical Interview for the DSM-IV (SCID-IV)
  3. Have persistent positive and negative symptoms despite having trialled, or being currently medicated, with antipsychotic medication; and
  4. are between the ages of 18 and 65.
* Concomitant medications including:

  1. Benzodiazepines,
  2. Mood stabilizers (lithium, valproic acid)
  3. Antidepressants (including serotonin reuptake inhibitors and tricyclic antidepressants) and anticholinergics will be allowed. Since carbamazepine has been shown to interfere with the effects of anodal tDCS, potential participants taking it will not be suitable for inclusion in the trial.
* Depression
* Participants will be included if they:

  1. Are competent to consent;
  2. Have a diagnosis of Major Depression and are currently experiencing a Major Depressive Episode as confirmed by the Structure Clinical Interview for the DSM-IV (SCID-IV);
  3. Are treatment resistant, defined as a failure to achieve a clinical response, or an inability to tolerate, an antidepressant trial of sufficient dose for at least 6 weeks; and
  4. Are between the ages of 18 and 75.
* Concomitant medications including:

  1. Benzodiazepines,
  2. Mood stabilizers (lithium, valproic acid)
  3. Antidepressants (including serotonin reuptake inhibitors and tricyclic antidepressants) and anticholinergics will be allowed. Since carbamazepine has been shown to interfere with the effects of anodal tDCS, potential participants taking it will not be suitable for inclusion in the trial.

Exclusion Criteria:

* Patients will be excluded if they:

  1. Have a DSM-IV history of substance abuse or dependence in the last 6 months;
  2. Have a concomitant major and unstable medical or neurologic illness;
  3. Are currently taking carbamazepine; or,
  4. Are pregnant.
* Patients will be withdrawn from the study if they:

  1. Withdraw consent;
  2. Experience significant clinical deterioration;
  3. Fail to tolerate the procedure; or,
  4. Develop a serious adverse event. In the event that a patient is withdrawn or drops out of the study, efforts will be made to obtain a final set of clinical, cognitive and neurophysiological measures at the time of withdrawal for a last observation carried forward analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Clinical Scales | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Fitzgerald, MBBS, MPM, PhD, FRANZCP, Principal Investigator — Alfred Psychiatry Research Centre
Locations (1):
- Alfred Psychiatry Research Centre, Prahran, Victoria, Australia